CLINICAL TRIAL: NCT05351164
Title: Evaluation of Safety and Efficiency of Metreleptin Treatment for Patients With Multiple Symmetric Lipomatosis (MSL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Amryt Pharma (Industry)
Responsible Party: Principal Investigator, Elif Oral, Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00206598
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Lipomatosis, Multiple Symmetrical
Keywords: Metreleptin
MeSH Terms: conditions — Lipomatosis, Multiple Symmetrical | interventions — metreleptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with MSL (Experimental)
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Study drug for injection is supplied in a carton containing 30 vials for reconstitution. Each vial contains 11.3 mg of the study drug as a sterile, white, solid, lyophilized cake or powder to deliver 5 mg/mL of the study drug when reconstituted with 2.2 mL of water for injection (WFI).

SUMMARY:
Participants (homozygous MFN2 [gene that provides instructions to produce the Mitofusin 2 protein] R707W) will be treated with Metreleptin, and effects on body composition, metabolic parameters and safety will be assessed over a 6 month intervention period. Additional safety will be assessed for 1 more year (up to 1.5 years total) in which adverse event data will be collected.

DETAILED DESCRIPTION:
In 2024, the IRB granted an amendment that allowed for continued data collection, including adverse events, up to 5 years per participant.

ELIGIBILITY:
Inclusion Criteria:

* Have the clinical diagnosis of MSL and being followed at University of Michigan (cohort to be studied in this proof-of-concept study is already available at Michigan).
* Willing and able to tolerate the study procedures.
* Willing and able to tolerate blood sampling.
* Having no condition that may impede successful data collection or interfere with testing parameters.
* <60 years of age.
* If female of childbearing potential:

  * Not breastfeeding.
  * Negative pregnancy test (human chorionic gonadotropin, beta subunit) at baseline.
* Can read, understand and sign approved informed consent form, communicate with study physician, and study team, and understand and comply with protocol requirements.

Exclusion Criteria:

* Presence of advanced liver disease (abnormal synthetic function, prothrombin time [PT], or albumin) in medical records
* Evidence of other etiologies of viral hepatitis in medical records
* Presence of active hematologic, bone marrow or other abnormalities that may increase risk of bleeding in medical records.
* Presence of HIV infection in medical records.
* Presence of End-stage renal disease (ESRD), active cancer, or >class 2 congestive heart failure based on medical history and physical examination.
* Active chronic infection (e.g., known chronic osteomyelitis or Tuberculosis [TB]). May have transient infections but must be free of active infection for two weeks prior to study visits.
* Unable to ambulate or tolerate trips to the University of Michigan Clinical Research Unit.
* Clinically relevant Coronary artery disease (CAD): history of stent or Coronary artery bypass graft surgery (CABG) with cardiologist confirmed angina.
* Presence of autoimmune disease.
* Hypersensitivity to metreleptin.
* General obesity not associated with congenital leptin deficiency.
* Any other condition that, in our opinion, may impede successful data collection.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2028-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elif Oral, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With MSL
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With MSL
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Truncal Adiposity
Description: A dual-energy X-ray absorptiometry (DEXA) scan was used to measure truncal adiposity at baseline and week 24. Truncal adiposity is the amount of fat a person has in the trunk area, and this outcome measure looked at the change in the fat in this area of the body in relation to the total fat in the participant's body. Results represent the change in the percentage of fat tissue from the trunk area to the total body.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: percentage of truncal body fat
Arm/Group | Patients With MSL
Number analyzed (Participants) | 4
percentage of truncal body fat
  Baseline | 22.8 (3.2)
  Week 24 | 16.0 (6.0)
Statistical Analysis 1: Comparison: Patients With MSL; Test type: Superiority; p = 0.004, t-test, 2 sided

2. Primary Outcome: Change in Total Adiposity
Description: A dual-energy X-ray absorptiometry (DEXA) scan was used to measure total adiposity at baseline and week 24. Total adiposity is the amount of fat participants had in the body compared to their total weight. Results represent the change in the percentage of fat tissue from the total body to the total weight.
Time Frame: Baseline, Week 24
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Patients With MSL
Number analyzed (Participants) | 4
percentage of body weight
  Baseline | 21.9 (2.3)
  Week 24 | 16.7 (4.7)
Statistical Analysis 1: Comparison: Patients With MSL; Test type: Superiority; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Patients With MSL
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With MSL (N=4)
fall from recreational vehicle (Injury, poisoning and procedural complications) | 1
weight loss (Metabolism and nutrition disorders) | 1
planned orthopedic surgery (Surgical and medical procedures) | 1
palpitations and chest discomfort (Cardiac disorders) | 1
Diarrhea or nausea (Gastrointestinal disorders) | 2
less stamina and strength (General disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Hematuria (self resolved) (Renal and urinary disorders) | 1
viral and non-serious bacterial infections (Infections and infestations) | 3
high blood pressure (Blood and lymphatic system disorders) | 1
high body temperature and intermittent shivering (General disorders) | 1
Chest discomfort and pain (Cardiac disorders) | 1
Syncope and collapse (General disorders) | 1
Nocturnal hunger (General disorders) | 1
Painful lipoma (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05351164/Prot_000.pdf